CLINICAL TRIAL: NCT04751981
Title: A Safety Trial for Evaluating Patient Specific Guides Accuracy for Pedicle Screw Insertion in Lumbar Fusion
Brief Title: Safety Trial of Patient Specific Guides for Lumbar Fusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10079
Record Dates: First submitted 2021-01-27; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Orthopedic Disorder of Spine
Keywords: Patient Specific Guides; Lumbar Fusion; Spine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Specific Guide (Experimental): Patients randomized into this group will have pedicle screws placed with the aid of patient specific surgical guides.
  Interventions: Procedure: Patient Specific Guide
- Navigation (Other): Patients randomized into this group will have pedicle screws placed with conventional navigation.
  Interventions: Procedure: Navigation

INTERVENTIONS:
Procedure: Patient Specific Guide — For lumbar fusion pedicle screws will be placed with the aid of patient specific guides.
  Arms: Patient Specific Guide
Procedure: Navigation — Conventional navigation will be used to place pedicle screws.
  Arms: Navigation

SUMMARY:
This is a single centre, non-blinded safety trial. Patients undergoing lumbar fusion will be treated using patient specific guides (PSG) or navigation. Patients requiring lumbar fusion will be treated using conventional surgical methods except when inserting pedicle screws, where half of the patients will be having screws inserted using PSGs. The conventional method of navigation and intraoperative imaging will be used in conjunction with PSGs, to confirm the safety of the guide trajectory. The primary outcome will be screw accuracy measured in degrees from planned trajectory and mm from the planned entry point.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Indication for lumbar spine surgery requiring pedicle screw instrumentation through a posterior approach with fusion.
* Recently has or requires a CT-scan of the spine
* No previous spine surgery on the level being used for patient specific guides
* Sufficient understanding of the English language or interpretation assistance available.

Exclusion Criteria:

* History of alcohol or drug abuse
* History of psychiatric disorders
* Previous spine surgery adjacent or at the level of the surgery
* Unable to read or comprehend the consent form/letter of information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Screw trajectory deviation | Day 1
  Measured as the angle in degrees deviated from the planned trajectory
Screw start point deviation | Day 1
  Measured as distance in millimeters from the planed start point.

SECONDARY OUTCOMES:
Pedicle Breach | Day 1
  Number, location and severity of any pedicle breaches
Adverse Event Rate & Serious Adverse Events | Day 1, Day 3, 6 weeks, 12 weeks, 26 weeks
  Measured intra-operatively and post-operatively
Guide Reliability | Day 1
  The reliability of patient specific guides will be measured as the number of cases that used the guides divided by the total number of cases in which guides were planned to be used.